CLINICAL TRIAL: NCT00006004
Title: A Randomized Phase II Trial of Paclitaxel-Carboplatin or Gemicitabine-Cisplatin in ECOG Performance Status 2 Non-Small Cell Lung Cancer Patients
Brief Title: Comparison of Two Combination Chemotherapy Regimens in Treating Non-small Cell Lung Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Eastern Cooperative Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: CDR0000068012; E-1599
Record Dates: First submitted 2000-07-05; First posted 2003-01-27 (Estimated); Last update posted 2023-06-15 (Actual); Status verified 2023-06

CONDITIONS: Lung Cancer
Keywords: recurrent non-small cell lung cancer; squamous cell lung cancer; large cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; adenocarcinoma of the lung; adenosquamous cell lung cancer; bronchoalveolar cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Carcinoma, Non-Small-Cell Lung; Adenocarcinoma of Lung; Adenocarcinoma, Bronchiolo-Alveolar | interventions — Carboplatin; Cisplatin; Gemcitabine; Paclitaxel

INTERVENTIONS:
Drug: carboplatin
Drug: cisplatin
Drug: gemcitabine hydrochloride
Drug: paclitaxel

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells. It is not yet known which combination chemotherapy regimen is more effective for treating non-small cell lung cancer.

PURPOSE: Randomized phase II trial to compare the effectiveness of two combination chemotherapy regimens in treating patients who have non-small cell lung cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

* Compare overall survival, response rate, and time to progression of patients with non-small cell lung cancer treated with paclitaxel and carboplatin versus gemcitabine and cisplatin.
* Compare the toxicities of each of these 2 regimens in this patient population.

OUTLINE: This is a randomized, multicenter study. Patients are stratified according to weight loss in the past 6 months (less than 5% vs at least 5%) and disease stage (stage IIIB with pleural or pericardial effusion or pleural implants vs stage IV/recurrent). Patients are randomized to one of two treatment arms.

* Arm I: Patients receive paclitaxel IV over 3 hours followed by carboplatin IV over 15-30 minutes on day 1.
* Arm II: Patients receive gemcitabine IV over 30 minutes on days 1 and 8 followed by cisplatin IV over 1 hour on day 1 only.

Treatment continues in both arms every 21 days for up to 6 courses in the absence of unacceptable toxicity or disease progression.

Patients are followed every 3 months for 2 years, every 6 months for 3 years, and then annually thereafter.

PROJECTED ACCRUAL: Approximately 40-90 patients (20-45 per arm) will be accrued for this study within 12 months.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically or cytologically confirmed non-small cell lung carcinoma of any of the following subtypes:

  * Squamous cell
  * Adenocarcinoma
  * Large cell anaplastic
  * Bronchioalveolar
  * Non-small cell carcinoma not otherwise specified
* No small cell anaplastic elements allowed
* Must have:

  * Recurrent disease after prior radiotherapy or surgery OR
  * Stage IV disease with distant metastases OR
  * Stage IIIB disease presenting with pleural or pericardial effusion on CT or chest x-ray or pleural implants documented pathologically or on CT or chest x-ray
* Bidimensionally measurable or evaluable disease
* Brain metastases allowed provided clinically stable after treatment with surgery and/or radiotherapy

PATIENT CHARACTERISTICS:

Age:

* 18 and over

Performance status:

* ECOG 2

Life expectancy:

* Not specified

Hematopoietic:

* Absolute neutrophil count at least 1,500/mm3
* Platelet count at least 100,000/mm3

Hepatic:

* Bilirubin no greater than 1.5 mg/dL
* SGOT no greater than 5 times upper limit of normal

Renal:

* Creatinine no greater than 1.5 mg/dL OR
* Creatinine clearance at least 60 mL/min

Cardiovascular:

* No uncontrolled high blood pressure, unstable angina, or congestive heart failure
* No myocardial infarction within the past 6 months
* No serious ventricular arrhythmias requiring medication

Other:

* Not pregnant or nursing
* Fertile patients must use effective contraception
* No other active malignancies requiring ongoing treatment
* No uncontrolled serious active infections
* No suspected hypersensitivity to agents that utilize Cremophor
* No evidence of neuropathy grade 2 or greater by history or physical examination

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* No prior chemotherapy for non-small cell lung cancer

Endocrine therapy:

* Not specified

Radiotherapy:

* See Disease Characteristics
* No prior radiotherapy to only site of measurable or evaluable disease unless subsequent progression documented by physical exam, radiograph, or pathology
* Recovered from prior radiotherapy
* No concurrent radiotherapy except for whole brain radiation for developing brain metastases

Surgery:

* See Disease Characteristics

Ages: 18 Years to 120 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Dates: Start 2000-08-22 (Actual); Primary Completion 2005-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Corey J. Langer, MD, Study Chair — Fox Chase Cancer Center
Locations (16):
- United States (13):
  - Emory University Hospital - Atlanta, Atlanta, Georgia
  - Iowa Methodist Medical Center, Des Moines, Iowa
  - Mercy Medical Center, Des Moines, Iowa
  - Iowa Lutheran Hospital, Des Moines, Iowa
  - Alegent Health-Midlands Community Hospital, Papillion, Nebraska
  - CCOP - Northern New Jersey, Hackensack, New Jersey
  - Cancer Institute of New Jersey, New Brunswick, New Jersey
  - MBCCOP - University of New Mexico HSC, Albuquerque, New Mexico
  - James P. Wilmot Cancer Center, Rochester, New York
  - CCOP - Oklahoma, Tulsa, Oklahoma
  - Milton S. Hershey Medical Center, Hershey, Pennsylvania
  - CCOP - Scott and White Hospital, Temple, Texas
  - CCOP - St. Vincent Hospital Cancer Center, Green Bay, Green Bay, Wisconsin
- Westmead Hospital, Westmead, New South Wales, Australia
- Instituto de Enfermedades Neoplasicas, Lima, Peru
- San Juan City Hospital, San Juan, Puerto Rico

REFERENCES:
- [Result] Langer C, Li S, Schiller J, Tester W, Rapoport BL, Johnson DH; Eastern Cooperative Oncology Group. Randomized phase II trial of paclitaxel plus carboplatin or gemcitabine plus cisplatin in Eastern Cooperative Oncology Group performance status 2 non-small-cell lung cancer patients: ECOG 1599. J Clin Oncol. 2007 Feb 1;25(4):418-23. doi: 10.1200/JCO.2005.04.9452. PMID 17264337
- [Result] Tester WJ, Stephenson P, Langer CJ, et al.: ECOG 1599: randomized phase II study of paclitaxel/carboplatin or gemcitabine/cisplatin in performance status (PS) 2 patients with advanced non-small cell lung cancer (NSCLC). [Abstract] J Clin Oncol 22 (Suppl 14): A-7055, 630s, 2004.
- [Result] Langer CJ, Stephenson P, Schiller J, et al.: ECOG 1599: randomized phase II study of paclitaxel/carboplatin vs cisplatin/gemcitabine in performance status (PS) 2 patients with treatment-naive advanced NSCLC. [Abstract] Lung Cancer 41 (Suppl 2): A-O52, S18, 2003.